CLINICAL TRIAL: NCT04454294
Title: Determining the Effect of Two Different Methods on Bleeding, Vital Signs and Oxygen Saturation in Children to Maintain Drain Patency After Cardiac Surgery
Brief Title: Determining the Effect of Two Different Methods in Children to Maintain Drain Patency After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2018/11
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Infant ALL; Congenital Heart Disease
Keywords: infant; congenital heart disease; drain patency; nursing
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): The first method; There is no application in maintaining the drain opening, but if there are necessary medical indications such as clot formation, blood accumulation in the drainage connections, lack of drainage, this group is intervened by milking method. In our study, this group will be taken as a control group, there will be a situation that requires intervention in the first 6 hours, and if the milking method is used, it will be excluded from the sample.
  Interventions: Other: Control
- Experimental Group (Absorption Group) (Experimental): The second method used to maintain the drain opening is the suction method. In this study, this group will be taken as the first experimental group. The suction method is a continuous use until the patient's drainage requirement and the physician's request is terminated by ensuring that the pressure is between 5 and 15 kPa (kilopascals) or 10-20 cm H20 after the appropriate negative pressure tracking system of the patient, who is accepted with intensive care under water drainage system, is established. system.
  Interventions: Other: Experimental Group (Absorption Group)
- Experimental Group (Milking Group) (Experimental): The third method is milking. In our study, this group will be taken as the 2nd experimental group. In the milking method, the process starts from the area close to the drain entry point. The latex tube is folded into 12 cm long pieces and gripped with two hands. The nurse repeats the process 3 times by compressing the parts gripped by the hand. This process is then used at intervals every hour to repeat the distal part.
  Interventions: Other: Experimental Group (Milking Group)

INTERVENTIONS:
Other: Control — Common Process Steps:
  1. Informed consent forms will be signed by those who wish to take part in the research.
  2. The form in which individual characteristics are questioned will be filled.
  3. Hands will be washed, gloves will be worn.
  4. Before the procedure, body temperature, heart rate, respiratory rate, blood pressure, oxygen saturation and bleeding amount will be recorded.
  5. Drains will be kept parallel to the ground and upright.
  6. Drainage hoses will not be bent and in-bed position will be provided in accordance with gravity.
  7. It will be ensured that all connections between the chest tubes and drainage unit are tight and secure.
  8. Dressings of the chest and mediastinum drains will be fixed on the patient's skin, so as not to interfere with drainage.
  9. To prevent the tubes from coming out, they will be fixed to the patient bed.
  Vital signs, Sp02 and bleeding amount will be recorded every hour for 6 hours after surgery
  Arms: Control
Other: Experimental Group (Absorption Group) — 1. Common process steps
  2. Appropriate negative pressure monitoring system of the patient, who is admitted to the intensive care unit with underwater drainage system, will be established.
     * The suction control room combined with the vacuum regulator will be filled with sterile distilled water up to the specified level (20 cm H2O).
     * From the vacuum regulator, the drain or drains will be connected tightly and by preventing the crimping, from the aspirator receptor hoses.
  3. Suction will begin with a low level and gradually increase the suction until a slight bubble is noticed in the suction control room.
  4. Suction pressure will be maintained between 5 and 15 kPa (kilopascals) or 10-20 cm H20.
  5. The application will continue without interruption until the patient's drain need and the doctor's request is ended.
  6. During the application, the patient's vital signs, Sp02 and bleeding amount will be recorded every hour without using an additional manipulation method.
  Arms: Experimental Group (Absorption Group)
Other: Experimental Group (Milking Group) — 1. Common process steps will be applied
  2. Operation will start from the area near the drain entrance point
  3. Latex tube will be folded into 12 cm long pieces and will be gripped with two hands
  4. The procedure will be repeated 3 times by compressing the parts gripped by the nurse hand.
  5. This process will be repeated in the distal part.
  6. After the application, the patient's vital signs, Sp02 and bleeding amount will be recorded every hour without using an additional manipulation method.
  Arms: Experimental Group (Milking Group)

SUMMARY:
In this study, it was aimed to determine the effect of the use of milking and sucking methods on bleeding amount, vital signs and oxygen saturation in children with chest and mediastinal drains after cardiac surgery.

DETAILED DESCRIPTION:
The patient admitted to the post-operative Cardiovascular Surgery Intensive Care Units primarily meets two nurses and is responsible for the arrangement of medical equipment, monitoring, monitoring, maintaining, recording, and performing the necessary treatments. Then the nurse positions the drain after checking the drain connections, checks the level of the drain and records it in the nurse follow-up note. Then, the method to be used in maintaining the drain opening is decided in cooperation with the physician.

Three different methods are currently used in the unit. The first method; There is no application in maintaining the drain opening, but if there are necessary medical indications such as clot formation, blood accumulation in the drainage connections, lack of drainage, this group is intervened by milking method. In our study, this group will be taken as a control group, there will be a situation that requires intervention in the first 6 hours, and if the milking method is used, it will be excluded from the sample.

The second method used to maintain the drain opening is the suction method. In this study, this group will be taken as the first experimental group. The suction method is a continuous use until the patient's drainage requirement and the physician's request is terminated by ensuring that the pressure is between 5 and 15 kPa (kilopascals) or 10-20 cm H20 after the appropriate negative pressure tracking system of the patient, who is accepted with intensive care under water drainage system, is established. system.

The third method is milking. In our study, this group will be taken as the 2nd experimental group. In the milking method, the process starts from the area close to the drain entry point. The latex tube is folded into 12 cm long pieces and gripped with two hands. The nurse repeats the process 3 times by compressing the parts gripped by the hand. This process is then used at intervals every hour to repeat the distal part.

After the applications related to the method to be used are performed, the patient's vital signs, Sp02 and bleeding amount are generally monitored every hour.

In this study, the data for each group will be collected before and after the procedure for 6 hours after surgery, from the moment the patient is admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

-Parents / legal guardian agree to participate in the study and sign the informed consent form,

* Having undergone congenital cardivascular surgery for the first time,
* Chest and / or mediastinal drain after cardiac surgery,
* Without secondary congenital anomaly and chronic disease,
* No neurological symptoms,
* No sepsis,
* 1 month - 1 year old age group,
* Anticoagulant use after surgery and during research,

Exclusion Criteria:

* Receiving extra corporal membrane oxygenation support,

  * Sternum admitted to open intensive care,
  * Receiving intraaortic balloon pump support,
  * Reoperative
* Complicated cases with bleeding diathesis and thought to be highly drained

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Body temperature | 6 hours after surgery
  This outcome will be considered as one of the vital signs. Body temperature measurement will be evaluated as axillary. The data for each group will be collected before and after the procedure for 6 hours after surgery
Heart rate | 6 hours after surgery
  This outcome will be considered as one of the vital signs. Heart rate measurement will be evaluated via monitor. The data for each group will be collected before and after the procedure for 6 hours after surgery
Respiratory rate | 6 hours after surgery
  This outcome will be considered as one of the vital signs. Heart rate measurement will be evaluated via monitor. The data for each group will be collected before and after the procedure for 6 hours after surgery
Blood pressure | 6 hours after surgery
  This outcome contains both systolic and diastolic blood pressure. Blood pressure measurement will be evaluated via monitor. The data for each group will be collected before and after the procedure for 6 hours after surgery
Oxygen saturation | 6 hours after surgery
  This outcome obtained with patient monitor. The data for each group will be collected before and after the procedure for 6 hours after surgery
Bleeding amount | 6 hours after surgery
  This outcome obtained with patient drain. The data for each group will be collected before and after the procedure for 6 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Ass. Prof., Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalli S, Saeed D, Fukamachi K, Gillinov AM, Cohn WE, Perrault LP, Boyle EM. Chest tube selection in cardiac and thoracic surgery: a survey of chest tube-related complications and their management. J Card Surg. 2009 Sep-Oct;24(5):503-9. doi: 10.1111/j.1540-8191.2009.00905.x. PMID 19740284
- [Background] Cook M, Idzior L, Bena JF, Albert NM. Nurse and patient factors that influence nursing time in chest tube management early after open heart surgery: A descriptive, correlational study. Intensive Crit Care Nurs. 2017 Oct;42:116-121. doi: 10.1016/j.iccn.2017.03.008. Epub 2017 Apr 28. PMID 28457690
- [Background] Lu C, Jin YH, Gao W, Shi YX, Xia X, Sun WX, Tang Q, Wang Y, Li G, Si J. Variation in nurse self-reported practice of managing chest tubes: A cross-sectional study. J Clin Nurs. 2018 Mar;27(5-6):e1013-e1021. doi: 10.1111/jocn.14127. Epub 2018 Feb 21. PMID 29076204
- [Background] Halm MA. To strip or not to strip? Physiological effects of chest tube manipulation. Am J Crit Care. 2007 Nov;16(6):609-12. No abstract available. PMID 17962505
- [Background] Sullivan B. Nursing management of patients with a chest drain. Br J Nurs. 2008 Mar 27-Apr 9;17(6):388-93. doi: 10.12968/bjon.2008.17.6.28906. PMID 18414310